CLINICAL TRIAL: NCT06619795
Title: Combined Effect of tDCS and Motor or Cognitive Activity in Patients With Alzheimer's Disease: A Proof-of-Concept Pilot Study
Brief Title: Combined Effect of tDCS and Motor or Cognitive Activity in Patients With Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was interrupted before reaching the planned sample size due to the SARS-CoV-2 pandemic.
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Valentina Varalta, Doctor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 140158
Record Dates: First submitted 2024-09-17; First posted 2024-10-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease (AD)
Keywords: Transcranial Direct Current Stimulation; Motor Activity; Cognitive Stimulation; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Motor Activity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CogS (Sham Comparator): The participants underwent cognitive treatment while receiving sham tDCS stimulation.
  Interventions: Device: Sham tDCS
- MotS (Sham Comparator): The participants underwent motor treatment while receiving sham tDCS stimulation
  Interventions: Device: Sham tDCS
- CogA (Experimental): The participants underwent cognitive treatment while simultaneously receiving anodal stimulation with tDCS.
  Interventions: Device: Anodal tDCS
- MotA (Experimental): The participants underwent motor treatment while simultaneously receiving anodal stimulation with tDCS.
  Interventions: Device: Anodal tDCS

INTERVENTIONS:
Device: Anodal tDCS — In addition to anodal tDCS stimulation, participants simultaneously underwent motor or cognitive therapy, depending on their assigned group.
  Arms: CogA; MotA
Device: Sham tDCS — In addition to Sham tDCS stimulation, participants simultaneously underwent motor or cognitive therapy, depending on their assigned group.
  Arms: CogS; MotS

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of combining tDCS with motor or cognitive activities on cognitive functions in patients with AD. Second aim is to investigate if tDCS has a different impact if it is combined with motor or cognitive activities.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Examination (MMSE) major or equal to 15;
* good level of compliance;
* acetylcholinesterase inhibitor treatment (e.g., donepezil, rivastigmine);
* no modifications of medication during the last four months.

Exclusion Criteria:

* behavioral disorders (e.g., aggressiveness);
* alcohol abuse;
* orthopedic pathology with risk of falls to the ground;
* respiratory pathology;
* severe auditory or visual deficits uncorrected;
* history of epileptic fits;
* anti-epileptic medication;
* metallic body implants; pacemaker;
* psychiatric, neurologic, systemic or metabolic disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) | From enrollment to the end of treatment at two weeks
  (Range: 0-30; higher score=best performance).

SECONDARY OUTCOMES:
Picture Recognition (PR) | From enrollment to the end of treatment at two weeks
  Picture Recognition (PR) is a subtest of the Rivermead Behavioral Memory Test-3, an ecological memory battery resembling everyday tasks, with the aim to measure daily memory function. The examinee is shown a set of picture and then is asked to recognize them from a further set of pictures at a later time in the testing session. It has two parallel version for monitoring changes over time (Range: 0-15; higher score=best performance).
Digit Span Test- Forward (DSF) | From enrollment to the end of treatment at two weeks
  Digit Span Test- Forward (DSF), used to measure span of immediate verbal recall. The examiner presents digits verbally at a rate of one per second. Examiner requires the participant to repeat the digits in the same order. The number of digits increases by one until the participant consecutively fails two trials of the same digit span length (higher score=best performance)
Digit Span Test- Backward (DSB) | From enrollment to the end of treatment at two weeks
  Digit Span Test- Backward (DSB), used to measure working memory. The examiner presents digits verbally and repeats the digits in reverse order. The number of digits increases by one until the participant consecutively fails two trials of the same digit span length (higher score=best performance).
Phonemic Fluency Test (PFT) | From enrollment to the end of treatment at two weeks
  Phonemic Fluency Test (PFT), used to measure processing speed, language production and executive functions. Participants are given one minute to produce as many unique words as possible starting with a given letter. The participant's score in each task is given by the number of correct words (higher score=best performance).
Visual Search Test (VST) | From enrollment to the end of treatment at two weeks
  Visual Search Test (VST), to assess visual-selective attention. Three matrices are shown to the subject and the patients has to cross in 45 minutes the target stimuli between distractors (Range: 0-60; higher score=best performance).
Sustained Attention to Response Test (SART) | From enrollment to the end of treatment at two weeks
  Sustained Attention to Response Test (SART): used to evaluate sustained attention and control inhibition. In the test, participants view a computer monitor on which a random series of single digits are presented at the regular rate of 1 per 1.15 seconds. The task is to press a single response key following each presentation with the exception of a nominated no-go digit, to which no response should be made. In the standard version of the test, 225 digits are presented in a continuous sequence over 4.3 minutes. The outcomes are false allarm (FA), omission (OM) and reaction times (RT) (higher score = worst performance)
Neuropsychiatric Inventory (NPI) | From enrollment to the end of treatment at two weeks
  Neuropsychiatric Inventory (NPI) to evaluate the presence, frequency and severity of behavioral disorders (Range 0-144; higher score = worst performance).

CONTACTS AND LOCATIONS:
Locations (1):
- Mons. A. Mazzali Foundation, Mantova, Italy

REFERENCES:
- [Derived] Fonte C, Rotundo G, Varalta V, Filosa A, Muti E, Barletta C, Evangelista E, Venturelli M, Picelli A, Smania N. Combined Effect of tDCS and Motor or Cognitive Activity in Patients with Alzheimer's Disease: A Proof-of-Concept Pilot Study. Brain Sci. 2024 Oct 30;14(11):1099. doi: 10.3390/brainsci14111099. PMID 39595863

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT06619795/Prot_SAP_000.pdf